CLINICAL TRIAL: NCT00694642
Title: Safety and Efficacy of Transendocardial Injection of Autologous Endothelial Progenitor Cell CD 133 for Therapeutics Angiogenesis
Brief Title: Safety and Efficacy of Autologous Endothelial Progenitor Cell CD 133 for Therapeutic Angiogenesis
Acronym: PROGENITOR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pilar Jimenez Quevedo (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor-Investigator, Pilar Jimenez Quevedo, MD, PhD, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: progenitorCD133
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Artery Disease; Refractory Angina
Keywords: Refractory angina
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- selected CD133+cells (Active Comparator): Transendocardial injection of selected CD133+cells
  Interventions: Biological: Selected CD 133+ cells
- no injection (No Intervention): Boths groups were treated with G-CSF, underwent an apheresis and NOGA mapping

INTERVENTIONS:
Biological: Selected CD 133+ cells — Endothelial progenitor cell CD 133
  Arms: selected CD133+cells

SUMMARY:
The purpose of this study is to determine whether transendocardial injections of autologous endothelial progenitor cells CD 133 is safe and feasible in patients with refractory angina.

DETAILED DESCRIPTION:
The PROGENITOR trial is a randomized, double-blinded, multicenter controlled trial including patients with Canadian cardiovascular society angina classification (CCS): II-IV and ischemic zones by SPECT but without any option for revascularization. Primary endpoint was to assess the safety and feasibility of transendocardial injection of selected CD133+cells. All patients were treated for 4-days with granulocyte colony-stimulating factor and underwent apheresis. CD133+ cells were selected with CliniMacs system and were injected transendocardially guided by the NOGA XP system.

ELIGIBILITY:
Inclusion Criteria:

* Functional class II- IV angina on maximal medical therapy
* Myocardial Ischemia/viability demonstrated by a reversible perfusion defect by means imaging techniques
* Patients should not be amenable to any type of revascularization procedure (percutaneous or surgical)
* Signed informed consent

Exclusion Criteria:

* Age <18 years or >75 years.
* Atrial fibrillation.
* LV thrombus
* Acute myocardial infarction in the last 3 months
* An LV wall thickness of <8 mm at the target site for cell injection
* A history of malignancy in the last 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac and cerebrovascular event | 6, 12 and 24 months
  cardiovascular death, non-fatal myocardial infarction (MI), ischemic stroke, need for revascularization or , procedure-related complications (: pericardial effusion/cardiac tamponade, vascular complications and sustained ventricular arrhythmias).

SECONDARY OUTCOMES:
Efficacy | 6 months
  The change in the myocardial perfusion defect at baseline versus follow-up measured by Single Photon Emission Computed Tomography (SPECT). Treadmill test, and clinical evaluation (CCS, nº angina episodes/month, nº nitroglycerin /month, Quality of life by seattle questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Jimenez-Quevedo, MD,PhD, Principal Investigator — Hostpial Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain